CLINICAL TRIAL: NCT05450029
Title: Neoadjuvant Chemoradiotherapy Plus Sintilimab for Intermediate/High Immunoscore Locally Advanced Rectal Cancer: A Single-Center, Open-Label, Single-Arm, Phase 2 Trial
Brief Title: Neoadjuvant Chemoradiotherapy Plus Sintilimab for Intermediate/High Immunoscore Locally Advanced Rectal Cancer
Acronym: SILAR
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yanhong Deng (Other)
Collaborators: GeneCast Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Yanhong Deng, Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIHSYSU-25
Record Dates: First submitted 2022-06-20; First posted 2022-07-08 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Rectal Cancer
Keywords: Rectal cancer; Immunoscore; MRD
MeSH Terms: conditions — Rectal Neoplasms | interventions — sintilimab; Chemoradiotherapy; Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chemoradiotherapy and PD1 inhibitor (Experimental): Chemoradiotherapy and PD1 inhibitor
  Interventions: Drug: Sintilimab

INTERVENTIONS:
Drug: Sintilimab — 6 cycles of mFOLFOX6 (oxaliplatin 85 mg/m2, and folinic acid 400 mg/m2 followed by bolus 5-fluorouracil 400 mg/m2 and 5-fluorouracil 2400mg/m2 as a 46-hour continuous infusion on day 1) followed by long course chemoradiotherapy (50 Gy in 25 fractions) followed by surgery. Patients will receive sintilimab 3mg/kg every 2 weeks during chemoradiotherapy (2nd-6th cycle).
  Other Names: Chemoradiotherapy and PD1 inhibitor

SUMMARY:
Immunoscore has been reported to be superior to microsatellite instability staging in predicting the disease-specific recurrence and survival for patients with colorectal cancer. However, the relationship between Immunoscore and its impact on patient's response to PD-1 blockade remains to be elucidated. This phase II, prospective, open label study is designed to evaluate the efficacy and safety of combination neoadjuvant chemoradiotherapy (nCRT) with the anti-PD-1 antibody sintilimab for intermediate/high Immunoscore locally advanced rectal cancer.

DETAILED DESCRIPTION:
This study investigates the safety, tolerability, and feasibility of sintilimab, an immunotherapy agent, in combination with nCRT for treatment of patients with intermediate/high Immunoscore locally advanced rectal cancer. Sintilimab is an anti-PD-1 inhibitor that works by enhancing the functional activity of the target immune cells to facilitate tumor regression and ultimately immune rejection.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years and ≤75 years.
2. Willing and able to provide written informed consent for participation in this study.
3. Treatment-naive patients with histological or cytological documentation of rectal adenocarcinoma (<12 cm from the anal verge).
4. Clinical stage of T3/T4 or N positive and M0, before nCRT.
5. Non complicated primary tumor (complete obstruction, perforation, bleeding).
6. Subjects with an intermediate or high immunoscore (according to Immunoscore®).
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
8. Women of childbearing potential who consent to practicing contraception during the period from giving informed consent to at least 23 weeks after the last dose of therapy.
9. Women of childbearing potential with a negative serum or urine pregnancy test within 24 hours prior to the start of study drug.
10. Subjects with normal organ and marrow function as defined below:

Leukocytes ≥ 3,000/k/uL; Absolute neutrophil count ≥ 1,500/k/uL; Platelet count ≥ 100,000/k/uL; Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN); AST (SGOT) ≤ 2.5 x institutional upper limit of normal (ULN); ALT (SGPT) ≤ 2.5 x institutional upper limit of normal (ULN); Serum creatinine ≤ 1.5 x institute upper limit of normal (ULN).

Exclusion Criteria:

1. Subjects with a history of a prior malignancy within the past 5 years, except for adequately treated basal cell or squamous cell skin cancer.
2. Subjects with a history of any arterial thrombotic event within the past 6 months. This includes angina (stable or unstable), myocardial infarction (MI), Transient Ischemic Attacks (TIA), or cerebralvascular accident (CVA).
3. Subjects with active lung disease (such as interstitial pneumonia, pneumonia, obstructive pulmonary disease, asthma) or active tuberculosis.
4. Subjects with any uncontrollable clinical problems, including but not limited to: active autoimmune disease, uncontrolled diabetes, uncontrolled hypertension, heart failure grade III/IV (NYHA-classification), or persistent or severe infection.
5. Subjects with a history of anti-PD-1, anti-PD-L1, or anti-PD-L2 therapy.
6. Subjects with known allergy to the study drugs or to any of its excipients.
7. Current or recent (within 4 weeks prior to starting study treatment) treatment of another investigational drug or participation in another investigational study.
8. Breast- feeding or pregnant women.
9. Subjects with significant unstable mental diseases or other medical diseases that may interfere with the safety of the subjects, obtaining informed consent, or compliance with the procedures for the clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response | 1 month after surgery
  Pathological complete response will be evaluated with American Joint Committee on Cancer (AJCC) Cancer Staging

SECONDARY OUTCOMES:
Margin-free (R0) resection rate | Immediately after the surgery
3-year event-free survival rate | 3 years after the surgery
3-year overall survival rate | 3 years after the surgery
Local recurrence | 3 years after the surgery
  Defined as an intrapelvic recurrence following a primary rectal cancer resection, with or without distal metastasis.
Tumor downstaging | during the 3-year period of follow-up
Tumor regression grade | during the 3-year period of follow-up
Number of participants with surgical complications | 30 days after surgery
Correlation between minimal residual disease (MRD) and survival | 3 years after the surgery
  The correlation between the status of MRD and the tumor local recurrence and metastasis.

CONTACTS AND LOCATIONS:
Overall Officials: Liang Kang, PhD,MD, Principal Investigator — Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- Department of colorectal surgery, the Sixth Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes